CLINICAL TRIAL: NCT00797862
Title: A Randomized, 32 Week Double-blind, Parallel-group, Multicenter Study to Compare the Efficacy and Safety of Initiating Treatment With Combination (Aliskiren/Amlodipine) Therapy in Comparison With the Sequential add-on Treatment Strategies in Patients With Essential Hypertension
Brief Title: Aliskiren and the Calcium Channel Blocker Amlodipine Combination as an Initial Treatment Strategy for Hypertension
Acronym: ACCELERATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CSPA100A2307
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Results first posted 2011-05-17 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension
Keywords: Aliskiren; Amlodipine; Hypertension; SPA1000; Norvasc
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Hydrochlorothiazide; aliskiren

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aliskiren + Amlodipine (Experimental): Eligible participants received oral aliskiren 150 mg + amlodipine 5 mg daily from week 1-8. From week 8 - 16, the dose of the combination treatment increased to aliskiren 300 mg + amlodipine 10 mg daily. From week 16-24, participants in this group continued combination treatment (aliskiren 300 mg + amlodipine 10 mg) for 8 weeks. At week 24, if blood pressure was not adequately controlled (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg) hydrochlorothiazide 12.5 mg was added to the combination (aliskiren 300 mg + amlodipine 10 mg) for an additional 8 weeks. Total treatment period =32 weeks.
  Interventions: Drug: Amlodipine; Drug: hydrochlorothiazide; Drug: Aliskiren
- Aliskiren Start - Amlodipine Add-On (Experimental): Eligible participants received oral aliskiren 150 mg daily from week 1-8. From week 8 - 16, the dose of aliskiren increased to 300 mg daily. From week 16-24, amlodipine 10 mg was added to the aliskiren 300 mg for 8 weeks (aliskiren 300 mg + amlodipine 10 mg). At week 24, if blood pressure was not adequately controlled (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg) hydrochlorothiazide 12.5 mg was added to the combination (aliskiren 300 mg + amlodipine 10 mg) for an additional 8 weeks. Total treatment period =32 weeks.
  Interventions: Drug: Amlodipine; Drug: hydrochlorothiazide; Drug: Aliskiren
- Amlodipine Start- Aliskiren Add-On (Experimental): Eligible participants received oral amlodipine 5 mg daily from week 1-8. From week 8 - 16, the dose of amlodipine increased to 10 mg daily. From week 16-24, aliskiren 300 mg was added to the amlodipine 10 mg for 8 weeks (amlodipine 10 mg + aliskiren 300 mg). At week 24, if blood pressure was not adequately controlled (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg) hydrochlorothiazide 12.5 mg was added to the combination (amlodipine 10 mg + aliskiren 300 mg) for an additional 8 weeks. Total treatment period =32 weeks.
  Interventions: Drug: Amlodipine; Drug: hydrochlorothiazide; Drug: Aliskiren

INTERVENTIONS:
Drug: Amlodipine — Amlodipine (5 mg and 10 mg) was provided as capsules taken orally once daily.
  Other Names: Norvasc
Drug: hydrochlorothiazide — Hydrochlorothiazide 12.5 mg capsules were taken orally once daily
  Other Names: Esidrix; HydroDIURIL; Oretic; Ezide; Hydro-Par
Drug: Aliskiren — Aliskiren 150 mg and aliskiren 300 mg were provided as film-coated tablets, taken orally once daily.
  Other Names: SPA 100

SUMMARY:
This study will compare the safety and efficacy of initial combination treatment with aliskiren + amlodipine to sequential add-on treatment strategies with aliskiren or amlodipine in patients with hypertension.

DETAILED DESCRIPTION:
This study was designed to evaluate if patients with hypertension treated early with a combination therapy would achieve better blood pressure (BP) control, than patients being treated with a classical sequential add-on therapy.

The study compared the effects of the two treatment strategies: Treatment initiation on a single compound, either with aliskiren or amlodipine, and then continuation with the combination of both versus treatment initiation with the combination of aliskiren/amlodipine and then continuation with the combination. The study also evaluated if the overall mean sitting systolic blood pressure (msSBP)-lowering effect during the study, as well as the change from baseline to study end in msSBP, are superior in the group having received combination therapy from the beginning.

The study further evaluated the BP-lowering efficacy and tolerability of both treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients ≥ 18 years of age
* Participants with essential hypertension:

  * Naive participants must have a mean sitting Systolic Blood Pressure (msSBP) ≥ 150 mmHg and < 180 mmHg at Visit 1 and Visit 2. (Participants are considered 'naïve' if they have never been treated with any antihypertensive medication.)
  * All participants must have a msSBP ≥ 150 mmHg and < 180 mmHg at Visit 2
* Written informed consent to participate in this study prior to any study procedures

Exclusion Criteria:

* Severe hypertension
* Pregnant or nursing (lactating) women
* Pre-menopausal women not taking accepted form of birth control
* Serum potassium ≥ 5.5 mEq/L (mmol/L) at Visit 1
* History of cardiovascular conditions
* Uncontrolled Type 1 or Type 2 diabetes mellitus
* Hypersensitivity to renin inhibitors, calcium channel blockers, or to drugs with similar chemical structures

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1254 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (10):
- Investigative Site, Toronto, Canada
- Investigative Site, San José, Costa Rica
- Investigative Site, Paris, France
- Investigative Site, Bonn, Germany
- Investigative Site, Athens, Greece
- Investigative Site, Guatemala City, Guatemala
- Investigative Site, Cape Town, South Africa
- Investigative Site, Basel, Switzerland
- Investigative Site, London, United Kingdom
- Investigative Site, Caracas, Venezuela

REFERENCES:
- [Derived] Brown MJ, Williams B, Morant SV, Webb DJ, Caulfield MJ, Cruickshank JK, Ford I, McInnes G, Sever P, Salsbury J, Mackenzie IS, Padmanabhan S, MacDonald TM; British Hypertension Society's Prevention and Treatment of Hypertension with Algorithm-based Therapy (PATHWAY) Studies Group. Effect of amiloride, or amiloride plus hydrochlorothiazide, versus hydrochlorothiazide on glucose tolerance and blood pressure (PATHWAY-3): a parallel-group, double-blind randomised phase 4 trial. Lancet Diabetes Endocrinol. 2016 Feb;4(2):136-47. doi: 10.1016/S2213-8587(15)00377-0. Epub 2015 Oct 18. PMID 26489809
- [Derived] Brown MJ, McInnes GT, Papst CC, Zhang J, MacDonald TM. Aliskiren and the calcium channel blocker amlodipine combination as an initial treatment strategy for hypertension control (ACCELERATE): a randomised, parallel-group trial. Lancet. 2011 Jan 22;377(9762):312-20. doi: 10.1016/S0140-6736(10)62003-X. Epub 2011 Jan 12. PMID 21236483

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A 2-4 week single-blind placebo run in. 7 patients were assigned a randomization number in error (3 each in the aliskiren/amlodipine initial treatment and aliskiren based add-on regimens and 1 in the amlodipine based add-on regimen). These patients did not take any double-blind study medication and were excluded from the Full Analysis Set (FAS).
Groups:
- Aliskiren+Amlodipine: Eligible participants received oral aliskiren 150 mg + amlodipine 5 mg daily from week 1-8. From week 8 - 16, the dose of the combination treatment increased to aliskiren 300 mg + amlodipine 10 mg daily. From week 16-24, participants in this group continued combination treatment (aliskiren 300 mg + amlodipine 10 mg) for 8 weeks. At week 24, if blood pressure was not adequately controlled (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg) hydrochlorothiazide 12.5 mg was added to the combination (aliskiren 300 mg + amlodipine 10 mg) for an additional 8 weeks. Total treatment period =32 weeks.
- Aliskiren Start-Amlodipine Add On: Eligible participants received oral aliskiren 150 mg daily from week 1-8. From week 8 - 16, the dose of aliskiren increased to 300 mg daily. From week 16-24, amlodipine 10 mg was added to the aliskiren 300 mg for 8 weeks (aliskiren 300 mg + amlodipine 10 mg). At week 24, if blood pressure was not adequately controlled (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg) hydrochlorothiazide 12.5 mg was added to the combination (aliskiren 300 mg + amlodipine 10 mg) for an additional 8 weeks. Total treatment period =32 weeks.
- Amlodipine Start-Aliskiren Add On: Eligible participants received oral amlodipine 5 mg daily from week 1-8. From week 8 - 16, the dose of amlodipine increased to 10 mg daily. From week 16-24, aliskiren 300 mg was added to the amlodipine 10 mg for 8 weeks (amlodipine 10 mg + aliskiren 300 mg). At week 24, if blood pressure was not adequately controlled (systolic blood pressure > 140 mmHg or diastolic blood pressure >90 mmHg) hydrochlorothiazide 12.5 mg was added to the combination (amlodipine 10 mg + aliskiren 300 mg) for an additional 8 weeks. Total treatment period =32 weeks.
Period: Overall Study
Arm/Group | Aliskiren+Amlodipine | Aliskiren Start-Amlodipine Add On | Amlodipine Start-Aliskiren Add On
Started | 620 (3 participants were mis-randomized and discontinued. Only 617 participants received study drug.) | 318 (3 participants were mis-randomized and discontinued. Only 315 participants received study drug.) | 316 (1 participant was mis-randomized and discontinued. Only 315 participants received study drug.)
Entered Double-Blind Treatment (FAS) | 617 | 315 | 315
Completed | 496 | 250 | 230
Not Completed | 124 | 68 | 86
Not completed — Adverse Event | 86 | 44 | 58
Not completed — Abnormal Test Procedure Result | 0 | 1 | 1
Not completed — Lack of Efficacy | 1 | 7 | 6
Not completed — No longer required study medication | 1 | 0 | 0
Not completed — Withdrawal by Subject | 14 | 7 | 7
Not completed — Lost to Follow-up | 11 | 0 | 5
Not completed — Administrative Problem | 4 | 0 | 0
Not completed — Protocol Violation | 4 | 6 | 8
Not completed — Mis-randomized | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren+Amlodipine | Aliskiren Start-Amlodipine Add On | Amlodipine Start-Aliskiren Add On | Total
Number analyzed (Participants) | 620 | 318 | 316 | 1254
Age Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.81) | 58.4 (10.83) | 58.1 (10.93) | 58.1 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 305 | 154 | 160 | 619
  Male | 315 | 164 | 156 | 635

OUTCOME MEASURES:

1. Primary Outcome: Overall Mean Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP) Over 8, 16 and 24 Weeks
Description: Systolic Blood Pressure was measured in a sitting position using a validated automated blood pressure monitor (the Omron device) according to Guidelines of the British Hypertension Society, at Baseline and over 8, 16 and 24 weeks of study treatment. The overall mean change in msSBP from baseline was estimated over three time points: Week 8, Week 16, and Week 24. Analysis used a repeated measures Analysis of Covariance (ANCOVA) model with treatment, visit, and region as factors, treatment by visit interaction and baseline msSBP as a covariate.
Time Frame: Baseline, 8 weeks, 16 weeks, and 24 weeks
Population: The analysis population included participants in the Full Analysis Set, (randomized participants who received at least one dose of study drug) for whom efficacy data was available for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren+Amlodipine | Aliskiren Start-Amlodipine Add On | Amlodipine Start-Aliskiren Add On
Number analyzed (Participants) | 604 | 312 | 313
mmHg | -25.34 (0.436) | -17.94 (0.600) | -19.81 (0.611)

2. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP) at Week 24
Description: Systolic Blood pressure was measured in a sitting position using a validated automated blood pressure monitor (the Omron device) according to Guidelines of the British Hypertension Society, at Baseline and 24 weeks of study treatment. Analysis used a repeated measures ANCOVA model with treatment, visit and region as factors, treatment by visit interaction and baseline msSBP as a covariate.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren+Amlodipine | Aliskiren Start-Amlodipine Add On | Amlodipine Start-Aliskiren Add On
Number analyzed (Participants) | 604 | 312 | 313
mmHg | -27.37 (0.546) | -26.34 (0.738) | -25.52 (0.782)

3. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP) at Week 32
Description: Diastolic Blood Pressure was measured in a sitting position using a validated automated blood pressure monitor (the Omron device) according to Guidelines of the British Hypertension Society, at Baseline and 32 weeks of study treatment. Change at Week 32 used a separate repeated measures ANCOVA model containing Week 8, 16, 24 and 32 data. Treatment, visit and region were factors in the model, treatment by visit interaction and baseline msDBP a covariate.
Time Frame: Baseline to 32 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren+Amlodipine | Aliskiren Start-Amlodipine Add On | Amlodipine Start-Aliskiren Add On
Number analyzed (Participants) | 604 | 312 | 313
mmHg | -12.96 (0.323) | -12.96 (0.446) | -11.62 (0.467)

4. Secondary Outcome: Overall Mean Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP) Over 8, 16, and 24 Weeks
Description: Diastolic Blood pressure was measured in a sitting position using a validated automated blood pressure monitor (the Omron device) according to Guidelines of the British Hypertension Society, at Baseline and over 8, 16 and 24 weeks of study treatment. The overall mean change in msDBP from baseline was estimated over three time points: Week 8, Week 16, and Week 24. Analysis used a repeated measures ANCOVA model with treatment, visit and regions as factors, treatment by visit interaction and baseline msDBP as a covariate.
Time Frame: Baseline, 8 weeks, 16 weeks and 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren+Amlodipine | Aliskiren Start-Amlodipine Add On | Amlodipine Start-Aliskiren Add On
Number analyzed (Participants) | 604 | 312 | 313
mmHg | -12.39 (0.247) | -8.37 (0.340) | -9.02 (0.347)

5. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP) at Week 24
Description: Diastolic Blood pressure was measured in a sitting position using a validated automated blood pressure monitor (the Omron device) according to Guidelines of the British Hypertension Society, at Baseline and 24 weeks of study treatment. Analysis used a repeated measures ANCOVA model with treatment, visit and region, as factors, treatment by visit interaction and baseline msDBP as a covariate.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren+Amlodipine | Aliskiren Start-Amlodipine Add On | Amlodipine Start-Aliskiren Add On
Number analyzed (Participants) | 604 | 312 | 313
mmHg | -13.64 (0.319) | -13.22 (0.431) | -12.25 (0.457)

6. Secondary Outcome: Percentage of Participants Achieving Overall Blood Pressure Control at 8, 16, 24 and 32 Weeks Endpoints
Description: Systolic & Diastolic Blood Pressure were measured in a sitting position using a validated automated blood pressure monitor (the Omron device) according to Guidelines of the British Hypertension Society, at Baseline and after 8, 16 , 24 and 32 weeks. Outcome is reported as percentage of participants achieving overall blood pressure control (msSBP <140 mmHg and msDBP <90 mmHg) at weeks 8, 16, 24 & 32 endpoints.
Time Frame: Baseline to week 8, 16, 24 and 32 endpoints
Population: The analysis population included participants in the Full Analysis Set, (randomized participants who received at least one dose of study drug) for whom efficacy data was available for this outcome measure. Last post-baseline observation was carried forward to each visit for the analysis of blood pressure control.
Measure: Number; unit: Percentage of Participants
Arm/Group | Aliskiren+Amlodipine | Aliskiren Start-Amlodipine Add On | Amlodipine Start-Aliskiren Add On
Number analyzed (Participants) | 604 | 312 | 313
Percentage of Participants
  Week 8 endpoint | 46.5 (0.566) | 22.8 (0.781) | 25.2 (0.816)
  Week 16 endpoint | 65.9 | 33.3 | 40.9
  Week 24 endpoint | 63.4 | 62.8 | 57.8
  Week 32 endpoint | 61.6 | 59.0 | 53.4

7. Post Hoc Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP) at Week 32
Description: Systolic Blood pressure was measured in a sitting position using a validated automated blood pressure monitor (the Omron device) according to Guidelines of the British Hypertension Society, at Baseline and 32 weeks of study treatment. Change at week 32 used a separate repeated measures ANCOVA model containing Week 8, 16, 24 & 32 data. Treatment, visit and region were factors in the model, treatment by visit interaction and baseline msSBP was a covariate.
Time Frame: Baseline to 32 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren+Amlodipine | Aliskiren Start-Amlodipine Add On | Amlodipine Start-Aliskiren Add On
Number analyzed (Participants) | 604 | 312 | 313
mmHg | -26.42 (0.566) | -25.75 (0.781) | -24.32 (0.816)

ADVERSE EVENTS:
Groups:
- Aliskiren: Eligible participants received oral aliskiren 150 mg daily from week 1-8. From week 8 - 16, the dose of aliskiren increased to 300 mg daily. From week 16-24, amlodipine 10 mg was added to the aliskiren 300 mg for 8 weeks (aliskiren 300 mg + amlodipine 10 mg). At week 24, if blood pressure was not adequately controlled (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg) hydrochlorothiazide 12.5 mg was added to the combination (aliskiren 300 mg + amlodipine 10 mg) for an additional 8 weeks. Total treatment period =32 weeks.
- Amlodipine: Eligible participants received oral amlodipine 5 mg daily from week 1-8. From week 8 - 16, the dose of amlodipine increased to 10 mg daily. From week 16-24, aliskiren 300 mg was added to the amlodipine 10 mg for 8 weeks (amlodipine 10 mg + aliskiren 300 mg). At week 24, if blood pressure was not adequately controlled (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg) hydrochlorothiazide 12.5 mg was added to the combination (amlodipine 10 mg + aliskiren 300 mg) for an additional 8 weeks. Total treatment period =32 weeks.
Arm/Group | Aliskiren + Amlodipine | Aliskiren | Amlodipine
Serious Adverse Events (participants affected / at risk) | 14/617 | 9/315 | 9/315
Other Adverse Events (participants affected / at risk) | 196/617 | 81/315 | 104/315
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren + Amlodipine (N=617) | Aliskiren (N=315) | Amlodipine (N=315)
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 0 | 0
Sigmoiditis (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1 | 0
Varicocele (Reproductive system and breast disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren + Amlodipine (N=617) | Aliskiren (N=315) | Amlodipine (N=315)
Oedema peripheral (General disorders) | 131 | 53 | 76
Joint swelling (Musculoskeletal and connective tissue disorders) | 46 | 20 | 21
Headache (Nervous system disorders) | 31 | 20 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with it's investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until publication of pooled data (i.e., data from all sites) in the clinical trial.